CLINICAL TRIAL: NCT07268586
Title: Intravenous Atropine in Reducing Reperfusion Arrhythmias, Conduction Abnormalities and Hypotension in Inferior ST-elevation Myocardial Infarction Undergoing Primary Percutaneous Coronary Intervention
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: FMASU R49/2025
Record Dates: First submitted 2025-11-01; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-10

CONDITIONS: Myocardial Infarction
Keywords: Atropine; Inferior ST elevation myocardial infarction
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Atropine arm (Active Comparator): This group will receive intravenous atropine 1 mg immediately before wire crossing
  Interventions: Drug: Intravenous atropine immediately before wire crossing during primary percutaneous coronary intervention
- Placebo arm (Placebo Comparator): This group will receive intravenous normal saline immediately before wire crossing
  Interventions: Drug: Intravenous normal saline as placebo immediately before wire crossing during primary percutaneous coronary intervention

INTERVENTIONS:
Drug: Intravenous atropine immediately before wire crossing during primary percutaneous coronary intervention — Intravenous atropine 1 mg immediately before wire crossing during primary percutaneous coronary intervention
  Arms: Atropine arm
Drug: Intravenous normal saline as placebo immediately before wire crossing during primary percutaneous coronary intervention — Intravenous normal saline as placebo immediately before wire crossing during primary percutaneous coronary intervention
  Arms: Placebo arm

SUMMARY:
People with acute inferior wall myocardial infarction will be given an intravenous drug called atropine that increases the heart rate to check if it prevents heart rhythm disturbances during performing coronary intervention

ELIGIBILITY:
Inclusion Criteria:

* Acute inferior ST elevation myocardial infarction

Exclusion Criteria:

* Execution of rescur percutaneous coronary intervention after thrombolysis
* Mechanical complications or no reflow or spontaneous reperfusion.
* Prior implantation of permanent or temporary pacemakers
* History of bradycardia, hypotension or ventricular tachycardia with a definitive cause (unrelated to the disease under study)
* Prior coronary artery bypass graft surgery
* Atropine contraindications Unwillingness to participate in the

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Conduction abnormalities | Periprocedurally
  Occurrence of conduction abnormalities
Reperfusion arrhythmias | Periprocedurally
  Occurrence of reperfusion arrhythmias

SECONDARY OUTCOMES:
Major adverse cardiac events | Periprocedurally
  Inhospital major adverse cardiac events including all-cause mortality, cardiovascular mortality, stroke and myocardial infarction

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Abbasia, Egypt

IPD SHARING:
Plan to Share IPD: No